CLINICAL TRIAL: NCT04256252
Title: Rituximab at Low dosE for neuromyelitiS optiCa spectrUm disordEr (RESCUE): a Prospective, Multicenter, Open-label, Follow-up Clinical Trial
Brief Title: Rituximab at Low dosE for neuromyelitiS optiCa spectrUm disordEr (RESCUE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Hongzeng Li, Principal investigator, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014TD-NMOSD
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; Rituximab
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab (Experimental): Intravenous rituximab was administered at a fixed dose of 100 mg once weekly for 3 weeks, followed by maintenance treatment with 100 mg rituximab every 6 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — A scheduled therapeutic regimen with low-dose rituximab was performed.
  Other Names: Rituxan

SUMMARY:
In this research, a prospective, multicenter(Tangdu Hospital of Fourth Military Medical University, Xi'an Gaoxin Hospital of Xi'an Medical College, Xianyang Central Hospital, Baoji Central Hospital, Xi'an Central Hospital, The First Hospital of Xi'an, The Fourth Hospital of Xi'an) open-label, follow-up clinical trial will carry out to evaluate the efficacy and safety of low-dose rituximab in treating NMOSD in Northwest China.

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD) is a group of autoimmune inflammatory demyelinating disease of the central nervous system primarily characterized with recurrent optic neuritis and longitudinally extensive transverse myelitis, leading to blindness and paralysis. Incremental disability due to clinical attacks make it essential to prevent relapses with immunosuppressive therapy. Since the serological pathogenic marker anti-aquaporin 4 immunoglobulin G (anti-AQP4 IgG) has been identified, NMOSD has unveiled its autoimmune features with close connections to B cell-mediated humoral immunity. Rituximab, a chimeric monoclonal antibody directly against human CD20 molecular on the surface of B cells, has been reported to deplete peripheral CD20+ B cells and to be highly effective for treating NMOSD, and therefore been recommended as first-line therapy for this disorder. Unfortunately, there are still no consensus statements on dosing and follow-up regimens, which needs investigations to explore the efficacy and safety of different rituximab strategies. Previous studies have provided pilot evidence supporting the use of low-dose rituximab in preventing relapses in Chinese patients with NMO/NMOSD, however, prospective multicenter studies are still needed to determine the effectiveness of the modified strategy in treating NMOSD.

ELIGIBILITY:
Inclusion Criteria:

Age between 16 and 75 years old;

Meet the 2007 or 2015 revised diagnostic criteria for NMOSD;

At least two relapses in recent two years and/or at least one attack or relapse in recent one years;

Expanded disability status scale (EDSS) score ≤7.0;

Willingness to sample collection, imaging study and other disease-related examinations and assessments;

Results of pregnancy tests for female patients with fertility during the screening period should be negative and effective contraception was used by the patient and her spouse during the study period;

Patients with informed consent.

Exclusion Criteria:

Other immunosuppressive agents are being used or have been discontinued for less than 3 months;

White blood cell count (WBC) <3 ×109/L, neutrophil count <1.5 ×109/L, hemoglobin (HGB) < 85 g/L, and platelet count (PLT) < 80×109/L;

Concomitant active liver disease or persistent elevation of transaminases more than three times above the normal upper limit;

Serious cardiovascular, kidney, blood and endocrine diseases, or history of malignant tumors, or severe infection;

Other chronic active immune diseases or stable conditions but requiring immunosuppressants or glucocorticoids, such as rheumatoid arthritis, scleroderma, Sjögren's syndrome, ulcerative colitis, AIDS, genetic or drug-induced immune deficiency;

Pregnant or lactating patients and those with family planning during the study period;

Allergy to rituximab and other components;

Inability to provide informed consent.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Annualized relapse rate at last follow-up visit | 12 months
  All the enrolled patients are followed up and annualized relapse rate is determined at last follow-up visit.

SECONDARY OUTCOMES:
Expanded disability status scale (EDSS) score at last follow-up visit | 12 months
  All the enrolled patients are followed up and expanded disability status scale (EDSS) score is determined at last follow-up visit. In general, the minimum and maximum scores of EDSS are 0 and 10, respectively, with higher scores meaning a worse outcome.
Rituximab-related adverse events | 1 month, 3 months, 6 months, 9 months, 12 months
  Rituximab-related adverse events (AEs) are evaluated and the rate of AEs is recorded.
Lesions in spinal cords | 6 months, 12 months
  Changes of lesions in spinal cord were evaluated by MRI scanning.
Circulating B cell monitoring | 6 months, 12 months
  Frequencies of total B cell (CD19+) and memory B cell (CD19+CD27+) in lymphocytes were assessed by flow cytometry.
Switch treatment | 6 months, 12 months
  Other immunosuppressive agents switched from rituximab and reasons for the switch are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzeng Li, Study Chair — Tang-Du Hospital